CLINICAL TRIAL: NCT06732882
Title: A Phase Ib, Multicentre, Randomised, Single-blind, Parallel-group, Placebo-controlled, Study to Characterise the Pharmacokinetics and Pharmacodynamics of AZD4604 Administered Via the Turbuhaler® Device in Adults With Mild Asthma
Brief Title: Study to Evaluate the Pharmacokinetics and Pharmacodynamics of AZD4604 Given Via the Turbuhaler® Device in Adults With Mild Asthma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8210C00006; 2024-516474-30-00 (Other: EU CT number)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: Turbuhaler device; Genuair device; Janus Kinase 1 inhibitor
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (5):
- AZD4604 dose A via Genuair (Experimental): Participants will receive dose A of AZD4604 via Genuair device twice daily
  Interventions: Drug: AZD4604; Device: Genuair
- AZD4604 dose A via Turbuhaler (Experimental): Participants will receive dose A of AZD4604 via Turbuhaler device twice daily
  Interventions: Drug: AZD4604; Device: Turbuhaler
- AZD4604 dose B via Turbuhaler (Experimental): Participants will receive dose B of AZD4604 via Turbuhaler device twice daily
  Interventions: Drug: AZD4604; Device: Turbuhaler
- Placebo via Genuair (Placebo Comparator): Participants will receive placebo via Genuair device twice daily
  Interventions: Other: Placebo; Device: Genuair
- Placebo via Turbuhaler (Placebo Comparator): Participants will receive placebo via Turbuhaler device twice daily
  Interventions: Other: Placebo; Device: Turbuhaler

INTERVENTIONS:
Drug: AZD4604 — Participants will receive AZD4604 via Genuair/Turbuhaler device.
  Arms: AZD4604 dose A via Genuair; AZD4604 dose A via Turbuhaler; AZD4604 dose B via Turbuhaler
Other: Placebo — Participants will receive placebo via Genuair/Turbuhaler device.
  Arms: Placebo via Genuair; Placebo via Turbuhaler
Device: Genuair — Participants will either receive AZD4604 or placebo via Genuair device.
  Arms: AZD4604 dose A via Genuair; Placebo via Genuair
Device: Turbuhaler — Participants will receive either AZD4604 or placebo via Turbuhaler device.
  Arms: AZD4604 dose A via Turbuhaler; AZD4604 dose B via Turbuhaler; Placebo via Turbuhaler

SUMMARY:
The study will investigate the Pharmacokinetic (PK), Pharmacodynamic (PD), the safety and tolerability of AZD4604, as well as to examine the effect of Fractional exhaled Nitric Oxide (FeNO) following the administration of the multiple doses of AZD4604 via Turbuhaler device.

DETAILED DESCRIPTION:
This is a multicentre, randomised, placebo-controlled, single-blind study to characterise PK and PD of AZD4604, administered twice daily (BID) using a Turbuhaler or a Genuair device.

Participants who have mild asthma with a raised FeNO will be randomised into the study to evaluate AZD4604 versus placebo, at 2 dose levels delivered via: a) the Turbuhaler device and b) the Genuair device.

The study will be comprised of:

* A screening period (Day -42 to Day-3)
* Participants will be randomised to one of 5 treatment arms where participants will either receive BID doses of AZD4604 or placebo from Day 1 to Day 9 and a single dose on Day 10.
* A follow-up Visit on Day 16

The total duration of the study will be for 58 days.

ELIGIBILITY:
Main Inclusion Criteria:

* Participant must be 18 to 65 years of age inclusive with suitable veins for cannulation or repeated venepuncture.
* Participants must have Physician-diagnosed mild asthma for at least 6 months prior to Screening Visit.
* ≥ 70% predicted for FEV1 at the Screening Visit AND on Day -1.
* Have a FeNO of ≥ 40 ppb at the Screening Visit and on Day -2.
* Body weight at least 50 kg and BMI within the range 18 to 35 kg/m2 (inclusive).
* Female participants must have a negative pregnancy test at the Screening Visit and on admission to the clinical site or prior to randomisation and must not be lactating. However, there are no restrictions on male participants or their female partners.
* Contraceptive use by females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed and dated informed consent prior to any study-specific procedure.

Main Exclusion Criteria:

* History of any clinically important disease or disorder which, in the opinion of the Principal Investigator (PI), may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History of cancer within the last 10 years (20 years for breast cancer) except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured. Any history of lymphoma is not allowed and disease history suggesting abnormal immune function.
* Participants with increased risk of infection.
* Have received any vaccine in the 30 days prior to the first dose.
* History or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of the study intervention.
* History of serious or severe adverse reaction or known hypersensitivity to AZD4604 or any of its additive constituents
* High sensitivity C-reactive protein > Upper Limit of Normal (ULN) at Screening Visit and Baseline/Run-in Period.
* Any clinically important abnormalities in clinical chemistry, haematology or urinalysis results as judged by the PI. The PI may consider appropriate ethnicity adjusted local reference ranges for haematology or clinical chemistry measurements, when available.
* Known or suspected history of drug abuse as judged by the PI and current smokers.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4604.
* Use of drugs with enzyme-inducing properties such as St John's wort within 3 weeks prior to the first administration of study intervention.
* History of alcohol abuse or excessive intake of alcohol as judged by the PI.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months prior to the Screening Visit.
* Participants who cannot communicate reliably with the PI or vulnerable participants.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting Electrocardiogram (ECG) and any clinically important abnormalities in the 12-lead ECG as considered by the investigator that may interfere with the interpretation of QTc interval changes.
* Female participants who are planning a pregnancy during the study period or within one month after the last dose of study intervention.
* Exacerbation of asthma symptoms within 6 months prior to Screening Visit and Day -1 requiring the use of oral, IM or IV steroids, antibiotics, accident and emergency visit, or hospital admission.
* If in the judgement of the PI, the participant has any ongoing or recent (ie, during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements, the participant should not be enrolled.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of study intervention in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Maximum observed drug concentration (Cmax) of AZD4604 | Day 9 (Pre-dose) and Day 10 (Pre-dose and Post-dose)
  The Cmax of AZD4604 at Day 10 of dosing with dose A and dose B when delivered by the Turbuhaler device will be characterised.
Time to reach maximum observed concentration (tmax) of AZD4604 | Day 9 (Pre-dose) and Day 10 (Pre-dose and Post-dose)
  The tmax of AZD4604 at Day 10 of dosing with dose A and dose B when delivered by the Turbuhaler device will be characterised.
Area under concentration-time curve in the dosing interval (AUCtau) of AZD4604 | Day 9 (Pre-dose) and Day 10 (Pre-dose and Post-dose)
  The AUCtau of AZD4604 at Day 10 of dosing with dose A and dose B when delivered by the Turbuhaler device will be characterised.
Apparent total body clearance (CL/F) of AZD4604 | Day 10 (Pre-dose and Post-dose)
  The CL/F of AZD4604 at Day 10 of dosing with dose A and dose B when delivered by the Turbuhaler device will be characterised.
Apparent volume of distribution based on the terminal phase (VZ/F) of AZD4604 | Day 10 (Pre-dose and Post-dose)
  The VZ/F of AZD4604 at Day 10 of dosing with dose A and dose B when delivered by the Turbuhaler device will be characterised.
Dose normalised AUCtau (AUCtau/D) of AZD4604 | Day 9 (Pre-dose) and Day 10 (Pre-dose and Post-dose)
  The AUCtau/D of AZD4604 at Day 10 of dosing with dose A and dose B when delivered by the Turbuhaler device will be characterised.
Dose normalised Cmax (Cmax/D) of AZD4604 | Day 9 (Pre-dose) and Day 10 (Pre-dose and Post-dose)
  The Cmax/D of AZD4604 at Day 10 of dosing with dose A and dose B when delivered by the Turbuhaler device will be characterised.

SECONDARY OUTCOMES:
Change from baseline to end of treatment in FeNO levels | From Screening visit (Day -42 to Day -3), Day -2 to Day 4, Day 9 to Day 10, Follow-up visit (Day 16)
  The change in FeNO levels from baseline to end of treatment after administration of AZD4604 delivered via Turbuhaler device will be evaluated.
Percentage of participants who achieve a FeNO < 25 ppb Cmax/D | From Screening visit (Day -42 to Day -3), Day -2 to Day 4, Day 9 to Day 10, Follow-up visit (Day 16)
  The percentage of participants who achieve a FeNO <25 ppb after administration of AZD4604 delivered via Turbuhaler device will be evaluated.
Change from baseline to end of treatment in FeNO levels | From Screening visit (Day -42 to Day -3), Day -2 to Day 4, Day 9 to Day 10, Follow-up visit (Day 16)
  The change in FeNO levels from baseline to end of treatment after administration of AZD4604 delivered via Turbuhaler and Genuair devices will be evaluated.
Maximum observed drug concentration (Cmax) of AZD4604 | Day 9 and Day 10
  The Cmax of AZD4604 at Day 10 of dosing with dose A, when delivered by the Genuair device will be characterised.
Time to reach maximum observed concentration (tmax) of AZD4604 | Day 9 and Day 10
  The tmax of AZD4604 at Day 10 of dosing with dose A, when delivered by the Genuair device will be characterised.
Area under concentration-time curve in the dosing interval (AUCtau) of AZD4604 | Day 9 and Day 10
  The AUCtau of AZD4604 at Day 10 of dosing with dose A, when delivered by the Genuair device will be characterised.
Apparent total body clearance (CL/F) of AZD4604 | Day 10
  The CL/F of AZD4604 at Day 10 of dosing with dose A, when delivered by the Genuair device will be characterised.
Apparent volume of distribution based on the terminal phase (VZ/F) | Day 10
  The VZ/F of AZD4604 at Day 10 of dosing with dose A, when delivered by the Genuair device will be characterised.
Dose normalised AUCtau (AUCtau/D) of AZD4604 | Day 9 and Day 10
  The AUCtau/D of AZD4604 at Day 10 of dosing with dose A, when delivered by the Genuair device will be characterised.
Dose normalised Cmax (Cmax/D) of AZD4604 | Day 9 and Day 10
  The Cmax/D of AZD4604 at Day 10 of dosing with dose A, when delivered by the Genuair device will be characterised.
Maximum observed drug concentration (Cmax) of AZD4604 | Day 9 and Day 10
  The Cmax of AZD4604 at Day 10 of dosing with dose A is compared via the Turbuhaler and Genuair devices.
Area under concentration-time curve in the dosing interval (AUCtau) | Day 9 and Day 10
  The AUCtau of AZD4604 at Day 10 of dosing with dose A is compared via the Turbuhaler and Genuair devices.

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (4):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Großhansdorf
  - Research Site, Lübeck
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, Harrow
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Wythenshawe

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/